CLINICAL TRIAL: NCT00704769
Title: Observational Study Evaluating the Safety and Efficacy of Desloratadine Syrup for Perennial Allergic Rhinitis in Indonesian Pediatric Patients
Brief Title: Response of Desloratadine Syrup in the Relief of Symptoms Associated With Perennial Allergic Rhinitis in Pediatric Patients (Study P04299)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P04299
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — desloratadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children with a history of perennial allergic rhinitis
  Interventions: Drug: Desloratadine (assigned by investigator as part of normal practice)

INTERVENTIONS:
Drug: Desloratadine (assigned by investigator as part of normal practice) — Desloratadine syrup, 2.5 mL (1.25mg) once daily for 2-5 year olds, 5 mL (2.5mg) once daily for 6-11 year olds, minimum 7 days of treatment, minimum of 2 visits
  Other Names: SCH 034117

SUMMARY:
Evaluate the safety and general clinical response of desloratadine syrup in the relief of symptoms associated with perennial allergic rhinitis in Indonesian pediatric patients.

DETAILED DESCRIPTION:
Children, ages 2-11, with a history of perennial allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Children patients of both sexes aged between 2-11 years, of either gender and any race
* Unequivocal history of perennial allergic rhinitis, including nasal congestion, sneezing, rhinorrhea, pruritus, and lacrimation
* Minimum score for inclusion: 10
* Capable of complying with the dosing regimen
* Free of any clinically significant disease (other than allergic rhinitis)
* Antihistamine must be justified by investigating doctor

Exclusion Criteria:

* Patients with asthma who require chronic use of inhaled or systemic corticosteroids
* History of frequent, clinically significant sinusitis or chronic purulent postnasal drip
* Patients with rhinitis medicamentosa
* History of hypersensitivity to desloratadine or any of its excipients
* Doctor deems unsuitable

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, ages 2-11, with a history of perennial allergic rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desloratadine
Started | 591
Completed | 591
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Desloratadine
Number analyzed (Participants) | 591
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 591
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.28 (2.92)
Sex/Gender, Customized [Number; unit: participants]
  Female | 238
  Male | 345
  Missing Information for sex | 8
Region of Enrollment [Number; unit: participants]
  Indonesia | 591

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: An adverse event was defined in the protocol to include any untoward medical occurrence or unfavorable and unintended sign in a subject administered a pharmaceutical product (at any dose). Additionally, any event that is associated with or observed in conjunction with a product overdose (whether accidental or intentional) or a product abuse and/or withdrawal were also considered an adverse event. The investigator assessed the relationship of any adverse event as either unlikely, possibly, or probably related to the use of study drug based on available information and protocol guidelines.
Time Frame: Minimum of 7 days after initiation of desloratadine
Measure: Number; unit: Participants
Arm/Group | Desloratadine
Number analyzed (Participants) | 591
Participants
  Nausea | 3
  Dizziness | 1

2. Primary Outcome: General Clinical Response of Desloratadine Syrup Based on the Physician's Judgments
Description: Physicians judged the subjects as good, excellent, fair, or poor.
Time Frame: Minimum of 7 days after initiation of desloratadine
Measure: Number; unit: Participants
Arm/Group | Desloratadine
Number analyzed (Participants) | 591
Participants
  Good | 350
  Excellent | 159
  Fair | 50
  Poor | 11

ADVERSE EVENTS:
Arm/Group | Desloratadine
Serious Adverse Events (participants affected / at risk) | 0/591
Other Adverse Events (participants affected / at risk) | 0/591

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other